CLINICAL TRIAL: NCT07348978
Title: Efficacy of Auricular Acupressure Combined With 0.1% Adapalene in the Treatment of Acne Vulgaris
Brief Title: Auricular Acupressure Combined With Adapalene for the Treatment of Acne Vulgaris
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Trang Le Thi Ha, Medical Doctor, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2464-DHYD-HDDD
Record Dates: First submitted 2025-12-26; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Acne Vulgaris
Keywords: Auricular Acupressure; Adapalene; Acne Treatment; Traditional Medicine; Complementary Therapy
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene; Gels

STUDY DESIGN:
Intervention Model Description: Participants were assigned to one of two parallel groups according to the study protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auricular Acupressure Plus Adapalene (Experimental): Participants received auricular acupressure combined with topical 0.1% adapalene.
  Interventions: Other: Auricular Acupressure; Drug: Adapalene 0.1% Gel
- Active Comparator (Experimental): Participants received topical 0.1% adapalene alone.
  Interventions: Drug: Adapalene 0.1% Gel

INTERVENTIONS:
Other: Auricular Acupressure — Auricular acupressure was performed by applying pressure to specific auricular points according to traditional medicine principles. The intervention was administered as an adjunctive therapy in combination with topical adapalene.
  Other Names: Ear Acupressure
  Arms: Auricular Acupressure Plus Adapalene
Drug: Adapalene 0.1% Gel — Topical adapalene 0.1% was applied to affected areas once daily as standard treatment for acne vulgaris.

SUMMARY:
Acne vulgaris is a common chronic inflammatory skin condition that can significantly affect quality of life. Standard treatments such as topical retinoids are effective but may not fully control symptoms in all patients.

This study evaluated the effectiveness of auricular acupressure combined with topical 0.1% adapalene compared with topical 0.1% adapalene alone in patients with acne vulgaris. Auricular acupressure is a non-invasive traditional medicine technique that may help regulate inflammatory responses and improve skin conditions.

The objective of this study was to determine whether the combination therapy provides greater improvement in acne severity and clinical outcomes than standard topical treatment alone.

DETAILED DESCRIPTION:
Acne vulgaris is a multifactorial inflammatory skin disease commonly affecting adolescents and young adults. Although topical retinoids such as adapalene are widely used and effective, some patients experience incomplete responses or persistent symptoms.

Auricular acupressure is a traditional therapeutic method that involves stimulating specific points on the ear and has been used to support systemic regulation and inflammatory control. This study was designed to explore the potential added benefit of auricular acupressure when combined with standard topical adapalene therapy.

This interventional study compared two treatment approaches in patients with acne vulgaris: auricular acupressure combined with topical 0.1% adapalene versus topical 0.1% adapalene alone. Participants were assigned to treatment groups according to the study protocol and followed for clinical assessment.

The primary objective of the study was to evaluate the effectiveness of the combination therapy in improving acne severity and overall clinical outcomes compared with standard treatment alone.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 to 35 years.
* Clinical diagnosis of mild to moderate acne vulgaris based on the Global Acne Grading System (GAGS).
* Willingness to comply with the study protocol and attend all scheduled visits.
* Provided written informed consent prior to participation.

Exclusion Criteria:

* Severe acne vulgaris requiring systemic treatment.
* Use of systemic acne treatments (such as isotretinoin, antibiotics, or hormonal therapy) within the past 4 weeks.
* Use of topical acne treatments within 2 weeks prior to enrollment.
* Presence of other dermatological conditions that may interfere with evaluation.
* Pregnancy or breastfeeding.
* Known allergy or hypersensitivity to adapalene or components of the intervention.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Change in Global Acne Grading System (GAGS) score | From baseline to week 4
  The Global Acne Grading System (GAGS) was used to assess acne severity. The total GAGS score was calculated at baseline and at the end of treatment. The primary outcome was the change in GAGS score from baseline to the end of treatment, and comparisons were made between the two study groups.

SECONDARY OUTCOMES:
Change in inflammatory and non-inflammatory acne lesion counts | From baseline to week 4
  The number of inflammatory lesions (papules and pustules) and non-inflammatory lesions (open and closed comedones) was recorded at baseline and weekly during treatment.
  The secondary outcome was the change in lesion counts from baseline to week 4 between the two treatment groups.
Change in Dermatology Life Quality Index (DLQI) score | From baseline to week 4
  Quality of life was assessed using the Dermatology Life Quality Index (DLQI), a validated questionnaire consisting of 10 items.
  The secondary outcome was the change in DLQI score from baseline to week 4, comparing the two study groups.
Incidence of treatment-related adverse events | During the 4-week treatment period
  Adverse events were monitored throughout the study period, including skin dryness, burning sensation, itching, erythema, and other local or systemic reactions.
  The frequency and type of adverse events were recorded and compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Bay Thi Nguyen, PhD, Principal Investigator — University of Medicine and Pharmacy at Ho Chi Minh City; Huy Chung Ly, Study Director — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (1):
- Le Van Thinh Hospital, Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical and privacy considerations and because the study was conducted at a single center